CLINICAL TRIAL: NCT04879849
Title: An Open-label, Phase 1, Dose-escalation Study to Evaluate the Safety and Preliminary Antitumor Activity of TAK-676 With Pembrolizumab Following Radiation Therapy in the Treatment of Non-small-cell Lung Cancer, Triple-negative Breast Cancer, or Squamous-cell Carcinoma of the Head and Neck That Has Progressed on Checkpoint Inhibitors
Brief Title: A Study of TAK-676 With Pembrolizumab After Radiation Therapy to Treat a Number of Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-676-1003; U1111-1252-0338 (Registry Identifier: WHO)
Record Dates: First submitted 2021-05-07; First posted 2021-05-10 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Dose Escalation Phase: Radiation + Pembrolizumab + TAK-676 (Experimental): Participants will receive image-guided radiation therapy between Day -8 and Day -2. Participants will then receive pembrolizumab 200 milligram (mg), infusion, intravenously (IV), once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by TAK-676 infusion with escalating doses (0.2 mg and above), IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurs first.
  Interventions: Drug: Pembrolizumab; Drug: TAK-676; Radiation: Image-guided radiation therapy

INTERVENTIONS:
Drug: Pembrolizumab — IV infusion.
Drug: TAK-676 — IV infusion.
Radiation: Image-guided radiation therapy — Radiation therapy.

SUMMARY:
In this study, adults with non-small-cell lung cancer (NSCLC), triple-negative breast cancer (TNBC) and squamous-cell carcinoma of the head and neck (SCCHN) will be treated with TAK-676 and pembrolizumab following radiotherapy. The main aims of this study are to check if people are improving after treatment with TAK-676, getting side effects from these combined treatments, and how much TAK-676 people with these cancers can receive without getting unacceptable side effects from it.

Participants will receive radiotherapy, then at least 40 hours later will receive pembrolizumab followed by TAK-676 slowly through a vein (infusion). Participants will receive an infusion of pembrolizumab at the same dose every 3 weeks. Different small groups of participants will receive lower to higher doses of TAK-676 on specific days of a 21-day cycle. This study will be happening at sites in North America.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-676. This study will evaluate the safety, tolerability and preliminary antitumor activity of TAK-676 with pembrolizumab following radiation therapy in the treatment of advanced NSCLC, TNBC or SCCHN that has progressed on checkpoint inhibitors (CPIs) and will estimate the maximum tolerated dose (MTD) and determine the recommended phase 2 dose (RP2D) of this combination.

The study will enroll approximately 65 participants. Participants will be assigned to dose escalating cohorts based on Bayesian Optimal Interval (BOIN) design. The starting dose of TAK-676 will be 0.2 mg and the subsequent dosing will be initiated based on the available safety and tolerability data from the previous cohort.

This multi-center trial will be conducted in the United States. There will be many clinic visits. The number of visits will depend on the number of cycles of treatment. Participants will attend an end of treatment (EOT) visit 30 days after receiving their last dose of study drug or before the start of subsequent systemic anticancer therapy, whichever occurs first. They might continue to have check-ups every 12 weeks if they left the study for a reason apart from their cancer getting worse.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
2. Participants must have at least 2 measurable lesions (i.e. ≥10 mm longest diameter for extranodal lesions, ≥15 mm short axis for lymph nodes), with at least one inside and at least one other outside of the radiation field. The tumor outside the radiation field must be accessible for biopsy, and the participant must consent to tumor biopsy at screening and during treatment.
3. Participants must have pathologically confirmed (cytological diagnosis is adequate) advanced or metastatic NSCLC, TNBC, or SCCHN who have:

   * Received or been offered all established standard of care (SOC) treatment options for which they are eligible; and
   * Progressed on CPIs in a prior line of therapy.
4. Adequate bone marrow, renal and hepatic functions.
5. Left ventricular ejection fraction (LVEF) >50%, as measured by echocardiogram or multiple-gated acquisition (MUGA) scan within 4 weeks before receiving the first dose of study drug.
6. Clinically significant toxic effects of previous therapy have recovered to Grade 1 (per NCI CTCAE, V5.0) or baseline, except for alopecia, Grade 2 peripheral neuropathy, and/or autoimmune endocrinopathies with stable endocrine replacement therapy.

Exclusion Criteria:

1. History of any serious cardiac or cerebrovascular conditions in the last 6 months, including uncontrolled congestive heart disease, unstable angina, myocardial infarction, hypertension greater than or equal to (≥) 160/100 millimeter of mercury (mmHg) in spite of optimal therapy, cardiac arrhythmias, pericardial effusion, cardiomyopathy, or symptomatic stroke. Chronic, stable atrial fibrillation on stable anticoagulation therapy, including low molecular weight heparin, will be allowed.
2. History of brain metastasis unless:

   * Clinically stable, (that is, treatment completed ≥4 weeks prior) following prior surgery, whole-brain radiation, or stereotactic radiosurgery, AND
   * Off corticosteroids.
3. Known history of uncontrolled autoimmune disorders, human immunodeficiency virus (HIV) infection, or other relevant congenital or acquired immunodeficiencies.
4. Chronic, active hepatitis (example, participants with known hepatitis B surface antigen seropositive and/or detectable hepatitis C virus [HCV]-ribonucleic acid [RNA]).
5. Treatment with any investigational products and systemic anticancer drugs (including vascular endothelial growth factor (VEGF) inhibitors), within 14 days or 5 half-lives, whichever is shorter, before Cycle 1 Day 1 (C1D1) of study drugs.
6. Prior radiation to lesions chosen for biopsy or response assessment.
7. Prior radiation to lesions other than those chosen for radiation therapy or biopsy in the current protocol within 4 weeks of C1D1 of study drug(s).
8. Use of systemic corticosteroids or other immunosuppressive therapy, concurrently or within 7 days of start of radiation therapy, with the following exceptions:

   * Topical, intranasal, inhaled, ocular, intra-articular, and/or other nonsystemic corticosteroids.
   * Physiological doses of replacement steroid therapy (example, for adrenal insufficiency).
9. Receipt of live attenuated vaccine (example, tuberculosis Bacillus Calmette-guerin [BCG] vaccine, oral polio vaccine, measles, rotavirus, yellow fiver) within 28 days of C1D1 of study drug(s).
10. Recipients of allogeneic or autologous stem cell transplantation or organ transplantation.
11. Ongoing Grade ≥2 infection or participants with Grade ≥2 fever of malignant origin.
12. Fridericia's corrected QT interval (QTcF) >450 milliseconds (msec) (males) or >475 msec (females) on a 12-lead electrocardiogram (ECG) during the screening period.
13. Grade ≥2 hypotension (that is, hypotension for which nonurgent intervention is required) at screening or during C1D1 pre-dose assessment.
14. Oxygen saturation less than (<) 92% on room air at screening or during C1D1 predose assessment.
15. Use of medications that are known clinical organic anion transporting polypeptide 1B1 (OATP1B1) and/or OATP1B3 inhibitors, concurrently or within 14 days of C1D1 of study drugs.
16. Current smoker.
17. Vaping within 90 days of C1D1 of study drugs.
18. Current diagnosis of pneumonitis, interstitial lung disease, severe chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis, other restrictive lung diseases, acute pulmonary embolism, or Grade ≥2 pleural effusion or ascites not controlled by tap or requiring indwelling catheters.
19. Treated with other stimulator of interferon genes (STING) agonists/antagonist and toll-like receptors agonists within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - Cedars Sinai Medical Center, Duarte, California
  - University of Chicago, Chicago, Illinois
  - Laura And Isaac Perlmutter Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Cooper BT, Iams WT, Page DB, Yuan Y, Gerber NK, Luke JJ, Gibbs JP, Gregory RC, Wong KK, Deng J, Perera SA, Ding K, Roberts ER, Berger A, Christensen CL, Tong EX, Maldonado Lopez AE, Appleman VA, Leonard EJ, Parent A, Huang YC, Bay C, Li C, Lineberry N, Raizer J, Olson DJ, Chmura SJ. Phase 1b Study of Dazostinag plus Pembrolizumab after Hypofractionated Radiotherapy in Patients with Select Advanced Solid Tumors. Cancer Res Commun. 2025 Dec 1;5(12):2249-2263. doi: 10.1158/2767-9764.CRC-25-0566. PMID 41296842
- [Derived] Carideo Cunniff E, Sato Y, Mai D, Appleman VA, Iwasaki S, Kolev V, Matsuda A, Shi J, Mochizuki M, Yoshikawa M, Huang J, Shen L, Haridas S, Shinde V, Gemski C, Roberts ER, Ghasemi O, Bazzazi H, Menon S, Traore T, Shi P, Thelen TD, Conlon J, Abu-Yousif AO, Arendt C, Shaw MH, Okaniwa M. TAK-676: A Novel Stimulator of Interferon Genes (STING) Agonist Promoting Durable IFN-dependent Antitumor Immunity in Preclinical Studies. Cancer Res Commun. 2022 Jun 23;2(6):489-502. doi: 10.1158/2767-9764.CRC-21-0161. eCollection 2022 Jun. PMID 36923556
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/6099884f1f1122001e30a78e

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 09 September 2021 to 30 April 2024.
Pre-assignment Details: Participants with a diagnosis of non-small-cell lung cancer (NSCLC), triple-negative breast cancer (TNBC) or squamous-cell carcinoma of the head and neck (SCCHN) were enrolled to receive radiotherapy, pembrolizumab 200 milligram (mg), intravenous (IV) infusion and TAK-676 IV infusion.
Groups:
- Radiation + Pembrolizumab +Dazostinag 0.2 Milligrams (mg): Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.2 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab +Dazostinag 0.4 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.4 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab +Dazostinag 0.8 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.8 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab +Dazostinag 1.6 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 1.6 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab +Dazostinag 2.5 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 2.5 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab +Dazostinag 3.5 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 3.5 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab +Dazostinag 5.0 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 5.0 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Radiation Only: Participants received radiation therapy with daily image guidance using a fractionated dose of 8 gray (Gy) × 3.
Period: Overall Study
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 Milligrams (mg) | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only
Started | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Initiation of Another Systemic Anticancer Treatment | 3 | 1 | 2 | 0 | 1 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2
Not completed — Completion of Follow-up Period and Assessments | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 0
Not completed — Transfer to long term safety study, single-patient Investigational New Drug application, or similar | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Reason Not Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who received at least 1 dose of radiation.
Groups:
- Radiation + Pembrolizumab +Dazostinag 0.2 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.2 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or TAK-676 or withdrawal of consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only | Total
Number analyzed (Participants) | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.50) | 65.5 (6.36) | 55.0 (9.20) | 59.7 (11.06) | 66.3 (16.18) | 62.0 (12.38) | 56.8 (10.70) | 73.0 (7.07) | 60.4 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 2 | 3 | 4 | 3 | 0 | 15
  Male | 2 | 2 | 3 | 1 | 4 | 2 | 3 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 4 | 3 | 7 | 5 | 5 | 2 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 5
  White | 3 | 2 | 3 | 1 | 6 | 4 | 3 | 2 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Based on TEAEs Severity
Description: AE: any untoward medical occurrence in participants administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. TEAE: any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug is considered treatment emergent. Severity grade is defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0. Grade 1: Mild (asymptomatic/mild symptoms; clinical/diagnostic observations only; intervention not indicated); Grade 2: Moderate (minimal, local/noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living [ADL]); Grade 3: Severe (severe/medically significant but not immediately life-threatening hospitalization/prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4: Life-threatening consequences, urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: From first dose of study drug administration up to 32 months
Population: Safety Analysis Set included participants who received at least 1 dose of radiation.
Measure: Count of Participants; unit: Participants
Groups:
- Radiation Only: Participants received radiation therapy with daily image guidance using a fractionated dose of 8 Gy × 3.
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only
Number analyzed (Participants) | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2
Participants
  Number of Participants Reporting one or More TEAEs | 4 | 2 | 4 | 3 | 7 | 5 | 6 | 2
  Number of Participants Reporting Any Grade 3 or Higher TEAEs | 0 | 1 | 4 | 1 | 3 | 2 | 4 | 1

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any TEAE that occurred during Cycle 1 and was considered by investigator to be at least possibly related to TAK-676 in combination with pembrolizumab. TEAEs meeting DLT definitions occurring in later cycles were considered in the determination of recommended phase 2 dose (RP2D) of TAK-676. DLTs were assessed based on NCI CTCAE version 5.0.
Time Frame: During Cycle 1 (cycle length= 21 days)
Population: The DLT-evaluable Analysis Set included participants who received all Cycle 1 doses of dazostinag, pembrolizumab and 3 doses of radiation without experiencing a DLT by the end of Cycle 1 follow-up and participants who received 3 doses of radiation, pembrolizumab, and the required dazostinag doses up until a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 7 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting One or More Treatment Emergent Serious Adverse Events (TESAEs)
Description: TEAE: any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug is considered treatment emergent. An SAE is defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is a medically important event that satisfies any of the following: a) may require intervention to prevent items 1 through 5 above. b) may expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization
Time Frame: From first dose of study drug administration up to 32 months
Population: Safety Analysis Set included participants who received at least 1 dose of radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only
Number analyzed (Participants) | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2
Participants | 0 | 1 | 3 | 1 | 3 | 0 | 3 | 1

4. Primary Outcome: Number of Participants With One or More TEAEs Leading to Dose Modifications
Description: TEAE: Any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug is considered treatment emergent.
Time Frame: From first dose of study drug administration up to 32 months
Population: Safety Analysis Set included participants who received at least 1 dose of radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only
Number analyzed (Participants) | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2
Participants | 2 | 1 | 3 | 0 | 4 | 3 | 4 | 1

5. Primary Outcome: Number of Participants With One or More TEAEs Leading to Treatment Discontinuation
Description: as for outcome 4
Time Frame: From first dose of study drug administration up to 32 months
Population: Safety Analysis Set included participants who received at least 1 dose of radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only
Number analyzed (Participants) | 4 | 2 | 4 | 3 | 7 | 6 | 6 | 2
Participants | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1

6. Secondary Outcome: Overall Response Rate (ORR) Assessed by Investigator as Per RECIST v1.1
Description: ORR was defined as the percentage of participants who achieved confirmed complete response (cCR) or confirmed partial response (cPR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version1.1 (RECIST, V1.1). Complete Response (CR) for Target Lesions was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 millimeter (mm) and for Nontarget Lesions was defined as disappearance of all nontarget lesions and normalization of tumor marker level and all lymph nodes must be non-pathological in size (<10 mm short axis). Partial Response (PR) was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest. Percentages were rounded off to nearest single decimal place.
Time Frame: Up to 32 months
Population: The response-evaluable analysis subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 4
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 14.3 [0.4 to 57.9] | 0 [0 to 0] | 25.0 [0.6 to 80.6]

7. Secondary Outcome: Duration of Response (DOR) For All Tumor Lesions Assessed by Investigator as Per RECIST v1.1
Description: DOR:time from 1st documentation of cPR/better to 1st documentation of progressive disease(PD) for responders(cPR or better).PR:at least 30% decrease in sum of LD of target lesions,with reference of baseline sum LD.2nd assessment confirming PR must have taken place at least 4 weeks after response of interest.PD of Target Lesions:at least 20% increase in sum of LD of target lesions,with reference of smallest sum LD recorded since treatment started/appearance of 1/more new lesions.PD of Nontarget Lesions:unequivocal progression of existing non-target lesions.Responders without documentation of PD were censored at last response assessment that was stable disease(SD) or better.SD:neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,with reference of smallest sum LD since treatment started.Evaluation was determined by investigator according to RECIST, V1.1.2nd assessment confirming CR/PR must have taken place at least 4 weeks after response of interest.
Time Frame: Up to 32 months
Population: The response-evaluable analysis subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Overall number of participants analyzed signifies participants who had cCR or cPR. Responders without documentation of PD were censored at the date of the last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
months |  |  |  |  | 9.26 [NA to NA] — 95% confidence interval (CI) was not estimable for a single participant. |  | NA [NA to NA] — All participants with a cCR or cPR within this arm group were right-censored for duration of response, thus estimates for median duration of response could not be calculated. Also, 95% CI was not estimable for a single participant.

8. Secondary Outcome: Time to Response (TTR) For All Tumor Lesions Assessed by Investigator as Per RECIST v1.1
Description: TTR was defined as the time from the date of first dose administration to the date of first documented cPR or better as determined by the investigator according to RECIST, V1.1. PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest.
Time Frame: Up to 32 months
Population: The Response-evaluable Analysis Subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Overall number of participants analyzed signifies participants who had cPR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
months |  |  |  |  | 1.38 [NA to NA] — 95% CI was not estimable for a single participant. |  | 5.39 [NA to NA] — 95% CI was not estimable for a single participant.

9. Secondary Outcome: Overall Response Rate Assessed by Investigator as Per Modified Intratumoral Immunotherapy RECIST (Modified itRECIST)
Description: ORR was defined as the percentage of participants who achieve cCR or cPR as determined by the investigator according to Modified itRECIST. CR for Target Lesions was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm and for Nontarget Lesions was defined as disappearance of all nontarget lesions and normalization of tumor marker level and all lymph nodes must be non-pathological in size (<10 mm short axis). PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 32 months
Population: The response-evaluable analysis subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 posttreatment evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 4
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 14.3 [0.4 to 57.9] | 0 [0 to 0] | 0 [0 to 0]

10. Secondary Outcome: Overall Response Rate For Tumors Within the Radiation Field (ORRirradiated)
Description: ORRirradiated was defined as the percentage of participants who achieve cCRirradiated or cPRirradiated in the tumor lesions lying within the radiation field as determined by the investigator according to modified itRECIST. CR for Target Lesions was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm and for Nontarget Lesions was defined as disappearance of all nontarget lesions and normalization of tumor marker level and all lymph nodes must be non-pathological in size (<10 mm short axis). PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 32 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 4
percentage of participants | 50.0 [1.3 to 98.7] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 14.3 [0.4 to 57.9] | 16.7 [0.4 to 64.1] | 0 [0 to 0]

11. Secondary Outcome: Overall Response Rate For Tumors Outside the Radiation Field (ORRnonirradiated)
Description: ORRnonirradiated was defined as the percentage of participants who achieve cCRnonirradiated or cPRnonirradiated in the tumor lesions lying outside of the radiation field as determined by the investigator according to modified itRECIST. CR for Target Lesions was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm and for Nontarget Lesions was defined as disappearance of all nontarget lesions and normalization of tumor marker level and all lymph nodes must be non-pathological in size (<10 mm short axis). PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 32 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 2 | 2 | 4 | 3 | 7 | 6 | 4
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 14.3 [0.4 to 57.9] | 0 [0 to 0] | 25.0 [0.6 to 80.6]

12. Secondary Outcome: Duration of Response (DOR) For Tumors Within the Radiation Field (DORirradiated)
Description: DORirradiated for tumor lesions lying within radiation field: as time from the date of first documentation of a cPRirradiated or better to the date of first documentation of irradiated PD in those lesions for irradiated responders (cPRirradiated or better). PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Irradiated responders without documentation of irradiated PD were censored at the date of last response assessment that is irradiated SD or better. PD of Target Lesions: at least a 20% increase in sum of the LD of target lesions, taking as reference the smallest sum LD recorded since treatment started or appearance of 1 or more new lesions. PD of Nontarget Lesions: unequivocal progression of existing non-target lesions. Evaluation was determined by the investigator according to modified itRECIST. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest.
Time Frame: Up to 32 months
Population: The Response-evaluable Analysis Subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Overall number of participants analyzed signifies participants who had cCRirradiated or cPRirradiated. Responders without documentation of PD were censored at the date of the last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1 | 0
months | NA [NA to NA] — All participants with a cCR or cPR within this arm group were right-censored for duration of response, thus estimates for median duration of response could not be calculated. Also, 95% CI was not estimable for a single participant. |  |  |  | NA [NA to NA] — All participants with a cCR or cPR within this arm group were right-censored for duration of response, thus estimates for median duration of response could not be calculated. Also, 95% CI was not estimable for a single participant. | NA [NA to NA] — All participants with a cCR or cPR within this arm group were right-censored for duration of response, thus estimates for median duration of response could not be calculated. Also, 95% CI was not estimable for a single participant. |

13. Secondary Outcome: Duration of Response (DOR) For Tumors Outside the Radiation Field (DORnonirradiated)
Description: DORnonirradiated for tumor lesions lying outside of the radiation field was defined as time from the date of first documentation of a cPRnonirradiated or better to the date of first documentation of nonirradiated PD in those lesions for nonirradiated responders (cPRnonirradiated or better). PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Nonirradiated responders without documentation of nonirradiated PD were censored at the date of last response assessment that is nonirradiated SD or better. Evaluation was determined by the investigator according to modified itRECIST. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest.
Time Frame: Up to 32 months
Population: The Response-evaluable Analysis Subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Overall number of participants analyzed signifies participants who had cCRnonirradiated or cPRnonirradiated. Responders without documentation of PD were censored at the date of the last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
months |  |  |  |  | NA [NA to NA] — All participants with a cCR or cPR within this arm group were right-censored for duration of response, thus estimates for median duration of response could not be calculated. Also, 95% CI was not estimable for a single participant. |  | NA [NA to NA] — All participants with a cCR or cPR within this arm group were right-censored for duration of response, thus estimates for median duration of response could not be calculated. Also, 95% CI was not estimable for a single participant.

14. Secondary Outcome: Time to Response (TTR) For Tumors Within the Radiation Field (TTRirradiated)
Description: TTRirradiated in the tumor lesions lying within the radiation field was defined as the time from the date of first dose administration to the date of first documented cPRirradiated or better as determined by the investigator according to modified itRECIST. PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest.
Time Frame: Up to 32 months
Population: The response-evaluable analysis subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Overall number of participants analyzed signifies participants who had cPRirradiated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1 | 0
months | 1.41 [NA to NA] — 95% CI was not estimable for a single participant. |  |  |  | 3.45 [NA to NA] — 95% CI was not estimable for a single participant. | 1.15 [NA to NA] — 95% CI was not estimable for a single participant. |

15. Secondary Outcome: Time to Response (TTR) For Tumors Outside the Radiation Field (TTR Nonirradiated)
Description: TTR nonirradiated in the tumor lesions lying outside of the radiation field was defined as the time from the date of first dose administration to the date of first documented cPRnonirradiated or better during the study in response-evaluable population as determined by the investigator according to modified itRECIST. PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. The second assessment confirming a CR or PR must have taken place at least 4 weeks after the response of interest.
Time Frame: Up to 32 months
Population: The Response-evaluable Analysis Subset, a subset of the comprehensive response-evaluable analysis set, included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Overall number of participants analyzed signifies participants who had cPRnonirradiated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
months |  |  |  |  | 1.38 [NA to NA] — 95% CI was not estimable for a single participant. |  | 5.39 [NA to NA] — 95% CI was not estimable for a single participant.

16. Secondary Outcome: Number of Participants With Increase in T-Cell Infiltration in Tumor Evaluated by Immunohistochemistry
Description: The T-cell infiltration levels were calculated as a change from pre-treatment to post-treatment levels. Number of participants who expressed increase in T-cell infiltration levels between the pre-treatment and post-treatment tumor biopsies are reported.
Time Frame: Up to approximately 32 months
Population: Overall number of participants analyzed are the participants who had paired samples (both pre-treatment and post-treatment biopsy sample) available for analysis, participants who did not have paired samples were not evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Radiation + Pembrolizumab +Dazostinag 0.2 mg | Radiation + Pembrolizumab +Dazostinag 0.4 mg | Radiation + Pembrolizumab +Dazostinag 0.8 mg | Radiation + Pembrolizumab +Dazostinag 1.6 mg | Radiation + Pembrolizumab +Dazostinag 2.5 mg | Radiation + Pembrolizumab +Dazostinag 3.5 mg | Radiation + Pembrolizumab +Dazostinag 5.0 mg | Radiation Only
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
participants |  |  |  | 1 |  |  | 1 |

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration up to 32 months
Description: Safety Analysis Set included participants who received at least 1 dose of radiation.
Groups:
- Radiation + Pembrolizumab + Dazostinag 0.2 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.2 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab + Dazostinag 0.4 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.4 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab + Dazostinag 0.8 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 0.8 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab + Dazostinag 1.6 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 1.6 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab + Dazostinag 2.5 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 2.5 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab + Dazostinag 3.5 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 3.5 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
- Radiation + Pembrolizumab + Dazostinag 5.0 mg: Participants received image-guided radiation therapy between Day -8 and Day -2. Participants then received pembrolizumab 200 mg, infusion, IV, once on Day 1 of Cycle 1 and then every 3 weeks in each 21-day treatment cycle, followed by dazostinag 5.0 mg infusion, IV, once on Days 1, 8, 15 in each 21-day treatment cycle until disease progression, intolerance to pembrolizumab or dazostinag or withdrawal of consent, whichever occurred first.
Arm/Group | Radiation + Pembrolizumab + Dazostinag 0.2 mg | Radiation + Pembrolizumab + Dazostinag 0.4 mg | Radiation + Pembrolizumab + Dazostinag 0.8 mg | Radiation + Pembrolizumab + Dazostinag 1.6 mg | Radiation + Pembrolizumab + Dazostinag 2.5 mg | Radiation + Pembrolizumab + Dazostinag 3.5 mg | Radiation + Pembrolizumab + Dazostinag 5.0 mg | Radiation Only
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 1/4 | 1/3 | 1/7 | 2/6 | 1/6 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2 | 3/4 | 1/3 | 3/7 | 0/6 | 3/6 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 4/4 | 3/3 | 7/7 | 5/6 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation + Pembrolizumab + Dazostinag 0.2 mg (N=4) | Radiation + Pembrolizumab + Dazostinag 0.4 mg (N=2) | Radiation + Pembrolizumab + Dazostinag 0.8 mg (N=4) | Radiation + Pembrolizumab + Dazostinag 1.6 mg (N=3) | Radiation + Pembrolizumab + Dazostinag 2.5 mg (N=7) | Radiation + Pembrolizumab + Dazostinag 3.5 mg (N=6) | Radiation + Pembrolizumab + Dazostinag 5.0 mg (N=6) | Radiation Only (N=2)
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Radiation + Pembrolizumab + Dazostinag 0.2 mg (N=4) | Radiation + Pembrolizumab + Dazostinag 0.4 mg (N=2) | Radiation + Pembrolizumab + Dazostinag 0.8 mg (N=4) | Radiation + Pembrolizumab + Dazostinag 1.6 mg (N=3) | Radiation + Pembrolizumab + Dazostinag 2.5 mg (N=7) | Radiation + Pembrolizumab + Dazostinag 3.5 mg (N=6) | Radiation + Pembrolizumab + Dazostinag 5.0 mg (N=6) | Radiation Only (N=2)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Fatigue (General disorders) | 1 | 1 | 3 | 1 | 5 | 3 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginitis gardnerella (Infections and infestations) | 0/2 | 0/0 | 0/1 | 0/2 | 0/3 | 1/4 | 0/3 | 0/0 — Number of participants at risk are female participants as this adverse event is specific to females.
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT04879849/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT04879849/SAP_001.pdf